CLINICAL TRIAL: NCT06796257
Title: A Retrospective Study on the Monaco-Serial Biological Function K-value Index Constraint for Cardiac Dose
Brief Title: Monaco-Serial Biological Function K-value Index Constraint for Cardiac Dose
Status: Not yet recruiting | Type: Observational
Sponsor: Jianjun Lai (Other)
Responsible Party: Sponsor-Investigator, Jianjun Lai, Advanced Medical Physicist, Zhejiang Hospital
Organization: Zhejiang Hospital (Other)
Other Study IDs: PDIBT002
Record Dates: First submitted 2025-01-19; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer Radiotherapy Planning
MeSH Terms: interventions — Radiotherapy Planning, Computer-Assisted

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — No Biospecimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: radiotherapy planning — In this study, CT localization images from 32 patients were retrospectively used for radiotherapy treatment planning. Three radiotherapy plans were designed based on different K-value intervals of the Monaco-Serial biological function constraint for the heart. The dose-volume parameters of the organs at risk were compared.

SUMMARY:
Breast cancer is the most common malignant tumor in women globally, with radiotherapy being a crucial adjunctive treatment . However, due to the proximity of the breast radiotherapy target to the heart, there is a dose-effect relationship between radiation dose and the risk of radiation-induced heart disease, leading to a significantly increased risk of cardiac complications in patients undergoing left-sided breast cancer radiotherapy . Modern radiotherapy planning systems, utilizing inverse intensity-modulated radiotherapy (IMRT) dose optimization algorithms, effectively limit radiation exposure to organs at risk while ensuring target dose conformity, and have been widely adopted in clinical practice . To further reduce heart dose, the deep inspiration breath-hold (DIBH) technique has become an essential method in recent breast cancer radiotherapy. DIBH increases lung volume, thereby expanding the distance between the target and the heart, enhancing dose attenuation in the target area and minimizing radiation exposure to the heart. The combination of DIBH with IMRT dose optimization algorithms effectively minimizes radiation to the heart and its substructures, reducing the risk of radiation-induced heart disease.

The Monaco radiotherapy planning system is one of the most widely used systems, employing the Monte Carlo dose calculation algorithm, which offers high accuracy and provides dose optimization results that are closer to actual radiation-induced damage. The Serial function within the system is one of the key biological optimization tools, particularly effective in dose constraints for the heart and its substructures. In Monaco-Serial, when the Power Law Exponent value, or K value, is set to 1, it is more sensitive to average dose constraints, and is commonly used for average dose constraints to the heart and its substructures in left breast cancer free-breathing IMRT (FB-IMRT) radiotherapy . However, in deep inspiration breath-hold IMRT (DIBH-IMRT), due to significant changes in the spatial relationship between the heart and the target, previous parameter settings may no longer provide the optimal solution, and there is currently no relevant research or To maximize the dose constraints for the heart and its substructures and reduce the risk of radiation-induced damage, this study conducted a retrospective analysis of 51 patients who had previously undergone left-sided breast cancer DIBH-IMRT. Radiotherapy plans were designed with different Monaco-Serial K values, followed by dosimetric comparisons. Additionally, the correlation between dose-volume changes of organs at risk (OARs) after K value adjustments and anatomical changes post-DIBH was analyzed. The aim is to identify the optimal K value setting for the Monaco-Serial biological optimization function in left-sided breast cancer DIBH-IMRT, providing data support for the clinical application of the Monaco system in designing DIBH-IMRT radiotherapy plans for left breast cancer.

The study included 51 left-sided breast cancer patients who underwent breast-conserving surgery followed by whole-breast radiotherapy, with an average age of 43.3 years (range: 29-72 years). All patients had good compliance and completed the entire DIBH treatment process. The workflow which includes CT simulation and positioning under both FB and DIBH, Monaco radiotherapy plan design, radiotherapy plan evaluation, and the correlation analysis of anatomical changes and dose reduction rates after DIBH.

ELIGIBILITY:
Inclusion Criteria:

* The patients who have successfully completed left-sided breast cancer DIBH-IMRT radiotherapy.

Exclusion Criteria:

* The patients who have not completed left-sided breast cancer DIBH-IMRT radiotherapy.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients who have successfully completed left-sided breast cancer DIBH-IMRT radiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2025-01-25 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
In the Monaco radiotherapy planning system, the dose-volume metrics for organs at risk and the metrics for changes in anatomical structures are extracted. | 2025.3.1
  In the radiotherapy planning system, the radiation dose-volume data for the patient's heart and lungs is extracted, specifically including the mean dose and maximum dose to the heart, the maximum dose and mean dose to the LAD (left anterior descending artery), and the V5, V20, V30, and mean dose to the affected lung tissue (units: Gy). Additionally, anatomical indicators following DIBH (Deep Inspiration Breath Hold) are observed in the radiotherapy planning system, including the volume increase of the affected lung (units: cm³ or %), the distance between the heart and the breast (units: cm), and the volume ratio between the heart and the affected lung (units: % or ratio).

IPD SHARING:
Plan to Share IPD: No